CLINICAL TRIAL: NCT03109782
Title: The Austrian Spinal Cord Injury Study (ASCIS)
Brief Title: The Austrian Spinal Cord Injury Study
Acronym: ASCIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Thomas Freude, Prof. M.D., Principal Investigator, Head of Traumatology, Paracelsus Medical University
Other Study IDs: ascis1411
Record Dates: First submitted 2017-03-31; First posted 2017-04-12 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Traumatic Spinal Cord Injury
Keywords: Spinal Cord Injury; Spine Surgery; Patient Registry; Trauma
MeSH Terms: conditions — Spinal Cord Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Traumatic spinal cord injury (tSCI) is a debilitating disease that leads to neurological deficits and often has long-term effects including severe lifelong disability. Given the devastating personal and economic consequences of SCI, it is critical to collect high-quality, prospective data. SCI has not been systemically assessed in Austria, and data regarding the etiology, incidence and prevalence are missing or significantly limited. More importantly to the individuals suffering from SCI, health care for SCI patients in Austria is not concentrated in specialized SCI centers but fragmented, which might result in a less effective recovery and rehabilitation of patients. Accordingly, the Paracelsus Medical University Salzburg (PMU) and the Austrian Social Insurance for Occupational Risks (AUVA) initiated the Austrian Spinal Cord Injury Study (ASCIS) at the beginning of 2012. ASCIS is defined as an organized network that uses observational methods to collect uniform longitudinal clinical data that can provide insight into current patient care parameters and evaluates the outcome of SCI patients. ASCIS was initiated with the aim to develop a registry for patients with tSCI in Austria as a base for addressing research questions, improving patient outcomes and establishing a platform for future clinical trials. Furthermore, a major goal of ASCIS is to get knowledge about the natural recovery after spinal cord lesion in a larger population of patients in the sense of a historical control group and bring new standardized assessment tools to the clinical setting. Due to the involvement of acute trauma hospitals and rehabilitation centers, ASCIS is uniquely positioned to capture detailed hospital-related information on the (very)-acute, rehabilitation and chronic phases of tSCI patients. Additionally, ASCIS is cooperation partner of the European Multi-Center Study about Spinal Cord Injury (EMSCI).

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from paresis or plegia after trauma
* First ASCIS assessment possible within the first 3 days after incidence
* Patient capable and willing of giving written informed consent
* No cognitive impairment which would preclude an informed consent (including severe traumatic brain injury)

Exclusion Criteria:

* Nontraumatic paresis or plegia (e.g. disc-herniation, tumor, AV-malformation, myelitis)
* Previously known dementia or severe reduction of intelligence, leading to reduced capabilities of cooperation or giving consent
* Peripheral nerve lesion above the level of lesion (e.g. Plexus brachialis impairment)
* Previously known polyneuropathy
* Severe craniocerebral injury

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care Centers
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-12 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in American Spinal Injury Association Impairment Scale (AIS) | Between day of trauma (0 day), 1-3 days, 14-40 days, 3 months, 6 months, 1 year and 2-3 years after injury

SECONDARY OUTCOMES:
Change in American Spinal Injury Association Motor Score (ASIAMS) | Between day of trauma (0 day), 1-3 days, 14-40 days, 3 months, 6 months, 1 year and 2-3 years after injury
Change in American Spinal Injury Association Sensory Score (ASIASS) | Between day of trauma (0 day), 1-3 days, 14-40 days, 3 months, 6 months, 1 year and 2-3 years after injury
Change in Spinal Cord Independency Measure (SCIM) | Between day of trauma (0 day), 1-3 days, 14-40 days, 3 months, 6 months, 1 year and 2-3 years after injury
Change in Walking Index for Spinal Cord Injury (WISCI II) | Between day of trauma (0 day), 1-3 days, 14-40 days, 3 months, 6 months, 1 year and 2-3 years after injury
Change in Timed Up and Go Test (TuG) | Between day of trauma (0 day), 1-3 days, 14-40 days, 3 months, 6 months, 1 year and 2-3 years after injury
Change in 6 Minute Walking Test (6MWT) | Between day of trauma (0 day), 1-3 days, 14-40 days, 3 months, 6 months, 1 year and 2-3 years after injury
Change in 10 Meter Timed Walk (10MTW) | Between day of trauma (0 day), 1-3 days, 14-40 days, 3 months, 6 months, 1 year and 2-3 years after injury
Change in quality of life using the Short Form 36 (SF-36) questionnaire | Between day of trauma (0 day), 1-3 days, 14-40 days, 3 months, 6 months, 1 year and 2-3 years after injury

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Resch, Prof. M.D., Study Chair — Paracelsus Medical University; Thomas Freude, Prof. M.D., Principal Investigator — University Clinic Salzburg, Department of Traumatology and Orthopaedics; Wolfgang Schaden, M.D. Dir., Study Director — Austrian Social Insurance for Occupational Risks (AUVA)
Locations (18):
- Austria (18):
  - Hospital Amstetten, Department of Traumatology, Amstetten
  - Ordensklinikum Barmherzige Brüder Eisenstadt, Department of Orthopaedic Surgery, Eisenstadt
  - Academic Hospital Feldkirch, Department for Trauma Surgery and Sports Traumatology, Feldkirch
  - Trauma Center Graz, Graz
  - University Clinic Graz, Department of Orthopaedics and Traumatology, Medical University Graz, Graz
  - Hospital Horn, Department of Traumatology, Horn
  - Hospital Klagenfurt, Department of Trauma Surgery and Sports Traumatology, Klagenfurt
  - Trauma Center Klagenfurt, Klagenfurt
  - Trauma Center Linz, Teaching Hospital of the Paracelsus Medical University Linz, Linz
  - University Clinic Linz, Department of Neurosurgery, Kepler University Linz, Linz
  - University Clinic Linz, Department of Orthopaedics and Traumatology, Kepler University Linz, Linz
  - Trauma Center Salzburg, Teaching Hospital of the Paracelsus Medical University Salzburg, Salzburg
  - University Clinic Salzburg, Department of Orthopaedics and Traumatology, Paracelsus Medical University, Salzburg
  - University Clinic St. Pölten, Department of Orthopaedics and Traumatology, Sankt Pölten
  - Lorenz Böhler Trauma Center Vienna, Vienna
  - SMZ Ost Donauspital, Department of Traumatology, Vienna
  - University Clinic Vienna, Department of Trauma Surgery, Medical University of Vienna, Vienna
  - Hospital Wiener Neustadt, Department of Traumaotlogy, Wiener Neustadt

REFERENCES:
- See also: Related Info — http://www.ascis.at/